CLINICAL TRIAL: NCT03513679
Title: Effect of Cervical Decompression Surgery on Neuromuscular Control and Kinematics During Gait in Adult Patients With Cervical Spondylotic Myelopathy
Brief Title: Gait in Adult Patients With Cervical Spondylotic Myelopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Texas Back Institute (Other)
Collaborators: Cervical Spine Research Society (Other)
Responsible Party: Principal Investigator, Ram Haddas, Director of Research, Texas Back Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TBIRF-CSRS
Record Dates: First submitted 2018-02-14; First posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Cervical Spondylotic Myelopathy
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Group (Experimental): Gait and balance testing as well as self-reported outcome assessments to be administered before and after surgery
  Interventions: Procedure: Surgical intervention
- Control Group (No Intervention): Gait and balance testing to be administered once in healthy subjects

INTERVENTIONS:
Procedure: Surgical intervention — Surgery to decompress the spinal cord, either with or without concurrent fusion
  Arms: Surgical Group

SUMMARY:
The purpose of this study is to evaluate the effect of cervical decompression surgery on the biomechanics of the lower extremities and spine during balance and gait in patients with cervical spondylotic myelopathy (CSM), before and after surgical intervention, and compare these parameters to an asymptomatic control group. To test our hypothesis that cervical decompression will improve preexisting gait disturbance, a gait analysis using dynamic surface EMG, video motion capture, and force plate analysis will be used. Patients 30 to 70 years old will be eligible for the study. Thirty subjects diagnosed with symptomatic CSM and are deemed appropriate surgical candidates, along with 30 healthy subjects with no spine pathology, will be enrolled in this study. Exclusion criteria include any history of previous lumbar/thoracic surgery or lower extremity surgery, BMI greater than 35, or currently pregnant. Each subject from the surgical group will be evaluated on 3 different occasions: 1) 1 week before surgery, 2) 3 months postoperative, and 3) 12 months postoperative. Control subject will only be evaluated once. Bilateral trunk and lower extremity neuromuscular activity will be measured during a full gait cycle using dynamic surface EMG measurements. Human video motion capture cameras will collect lumbar spine and lower and upper extremity joint angles. Ground reaction forces (GRFs) will be collected from a 5 foot stretch of force platforms in order to define a full gait cycle.

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM) is a neurologic condition resulting from spinal cord compression caused by degenerative narrowing of the cervical spinal canal. CSM is most common after the age of 50 years, but the age of onset is variable depending on the degree of congenital spinal canal narrowing. Progressive degenerative changes in the cervical spine, such as disc bulges or herniations, facet hypertrophy, ligamentum flavum thickening, and degenerative vertebral spondylolisthesis, can all contribute to progressive spinal cord compression. The end result is chronic compression of the spinal cord and/or nerve roots leading to impaired blood flow, which can result in frank damage within the spinal cord itself. CSM is characterized by a wide variety of clinical presentations, which can include neck pain, numbness or weakness in the extremities, hand clumsiness, and, classically, gait disturbances. This typically manifests as difficulty with balance, but patients with more advanced myelopathy can also develop a stiff, spastic gait.

Surgical treatment of CSM revolves around decompressing the spinal cord, either with or without concurrent fusion. Many surgical strategies have been proposed. Anterior surgical approaches include anterior cervical discectomy and fusion or anterior corpectomy and fusion. Posterior surgical approaches include laminectomy with or without fusion, or laminoplasty. The choice of surgical approach is specific to each patient based upon the extent and location of the pathology, the presence or absence of deformity or spinal instability, the sagittal alignment of the spine, the presence or absence of ossification of the posterior longitudinal ligament (OPLL), as well as other patient co-morbidity factors and surgeon preference. While there may be some debate as to when patients with radiographic cervical stenosis should undergo decompressive surgery, most surgeons would agree on surgery for patients with moderate or severe clinical myelopathy.

Altered gait is frequently seen with CSM, and has been reported to be improved by surgical intervention. A stiff or spastic gait is also characteristic of CSM in its later stages. Many clinical studies have determined that patients with CSM have a slower gait speed, prolonged double support duration, and reduced cadence compared to healthy controls.Previous studies also identified reduced knee flexion during swing in the early stages of the disease, and, in more severe cases, decreased ankle plantar flexion at the terminal stance and reduced knee flexion during loading response.

Upright stance and body stability depends on the vestibular, visual, and somatosensory systems.These systems contribute to the maintenance of postural control. The spinal cord, particularly the dorsal column, is an integral part of the somatosensory system.The dorsal columns relay the position and vibration sensations as well as play an important role in maintaining postural stability and conveying sensory information such as deep sensations to the lower limbs.When the dorsal column of the spinal cord is compressed, the functions of vibration sense, deep sensibility, and joint position sense are lost. CSM patients were found to have impaired knee proprioception when using electrogoniometer.22 A damaged spinal cord causes impaired body balance because of proprioceptive loss, and patients develop ataxia in the lower limbs.

Jean Dubousset, first introduced the concept of the cone of economy and balance (COE) in 1994. The COE refers to a stable region of standing posture. The fundamental assumption is that swaying outside one's individual cone challenges the balance mechanisms and expends critical energy. Balance is defined as the ability of the human body to maintain its center of mass within the base of support with minimal postural sway. Sway is the movement of the COM in the horizontal plane when a person is standing in a static position. Balance efficiency is defined as the ability of the patients to maintain their COM within the COE with minimal sway and energy expenditure.Maintenance of balance requires coordination between the sensorineural and musculoskeletal systems. Very few studies have looked at functional balance in CSM patients. These studies used a stabilometer to measure center of gravity. During a 30 seconds balance test with closed eyes, CSM patients swayed significantly more and had greater postural instability compared to healthy controls. Neither of those studies reported on neuromuscular activity during a functional balance test. Haddas et al.was first to introduce a method to objectively quantify the COE and neuromuscular energy expenditure during a dynamic balance test.

There is very little literature investigating the effect of surgical intervention on a CSM patient's balance and gait using human motion analysis both before and after surgery. In fact, there have not been any studies examining how surgical intervention for CSM can improve patients' balance and gait utilizing objective neuromuscular data as well as full body kinematic analysis. Additionally, none of the previous studies have been able to validate self-reported pain and functional outcome measures utilizing a human motion capture system and EMG.

This study explores the effect of CSM on human balance and gait and will utilize kinematic balance and gait analyses to examine the dynamic range of motion of the spine and lower extremities, along with neuromuscular data from surface EMG to precisely define the timing and degree of spine and lower extremity muscle activation and peak activity, as well as measurements of ground reaction forces throughout the gait cycle. All of this will be compared pre- and post-operatively and also with a healthy control group in order to determine the extent to which CSM affects the biomechanics of and neuromuscular control during balance and gait and how this changes after surgical intervention. We will also be able to correlate these objective measures with patient self-reported pain and function based on commonly used outcome instruments.

In summary, the purpose of this study is to explore the level of functional compromise, both objectively and with patient-reported outcome measures, in patients with CSM and to quantify the possible benefit of surgical intervention on the biomechanics and neuromuscular control of the spine and lower extremities as evaluated by balance and gait analyses using dynamic EMG, video motion capture, force plate analysis, and validated patient-reported outcome metrics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 years and older
2. Diagnosis of CSM with correlative imaging studies (MRI or CT-myelogram)
3. Able to ambulate without assistance and stand without assistance with participant eyes open for a minimum of 10 seconds
4. Able and willing to attend and perform the activities described in the informed consent within the boundaries of the timelines set forth for pre-, and post-operative follow-up

Exclusion Criteria:

1. History of prior attempt at fusion (successful or not) at the indicated levels, (history of one level fusion is not an exclusion)
2. Major lower extremity surgery or previous injury that may affect gait (a successful total joint replacement is not an exclusion)
3. BMI higher than 35
4. Neurological disorder (beside cervical spondylotic myelopathy), diabetic neuropathy or other disease that impairs the patient's ability to ambulate or stand without assistance
5. Usage of blood thinners
6. Pregnant or wishing to become pregnant during the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Kinematic Variables Change assessed with human motion capture system | Baseline; 3 and 12 months after surgery
  3-Dimensional Range of Motion (ROM) during the stance and swing phase of the spine, pelvis, hip, knee, ankle, shoulder, and elbow joint angles along with CoM and head sway and displacement
Kinetic Variables Change assessed with human motion capture system | Baseline; 3 and 12 months after surgery
  Vertical Ground Reaction Forces (GRF)
Neuromuscular Variables Change assessed with an Electromyography | Baseline; 3 and 12 months after surgery
  Bilateral peak magnitude during the stance phase
Spatio-Temporal Variables Change assessed with human motion capture system | Baseline; 3 and 12 months after surgery
  Walking speed

SECONDARY OUTCOMES:
Patient Self-Reported Outcome Assessments Change | Baseline; 3 and 12 months after surgery
  Visual analog scale (VAS) for lower back pain, neck and arm pain, and leg pain. Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change | Baseline; 3 and 12 months after surgery
  Oswestry Disability Index (ODI, version 2.1.a). Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change | Baseline; 3 and 12 months after surgery
  Neck Disability Index (NDI). Scale range from 0 (no pain) - 10 (most pain)
Patient Self-Reported Outcome Assessments Change | Baseline; 3 and 12 months after surgery
  Modified Japanese Orthopaedic Association scale (mJOA). Scale range from 0 (no pain) - 18 (most pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Back Institute, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Portney LG, Watkins MP. Foundation of clinical research: applications to practiceed. Upper Saddle River, New Jersy: Julie Levin Alexander, 2009.
- [Result] Rhee JM, Heflin JA, Hamasaki T, Freedman B. Prevalence of physical signs in cervical myelopathy: a prospective, controlled study. Spine (Phila Pa 1976). 2009 Apr 20;34(9):890-5. doi: 10.1097/BRS.0b013e31819c944b. PMID 19352222
- [Result] Emery SE. Cervical spondylotic myelopathy: diagnosis and treatment. J Am Acad Orthop Surg. 2001 Nov-Dec;9(6):376-88. doi: 10.5435/00124635-200111000-00003. PMID 11767723
- [Result] Rao R. Neck pain, cervical radiculopathy, and cervical myelopathy: pathophysiology, natural history, and clinical evaluation. J Bone Joint Surg Am. 2002 Oct;84(10):1872-81. doi: 10.2106/00004623-200210000-00021. No abstract available. PMID 12377921
- [Result] Salvi FJ, Jones JC, Weigert BJ. The assessment of cervical myelopathy. Spine J. 2006 Nov-Dec;6(6 Suppl):182S-189S. doi: 10.1016/j.spinee.2006.05.006. PMID 17097537
- [Result] Eskander MS, Aubin ME, Drew JM, Eskander JP, Balsis SM, Eck J, Lapinsky AS, Connolly PJ. Is there a difference between simultaneous or staged decompressions for combined cervical and lumbar stenosis? J Spinal Disord Tech. 2011 Aug;24(6):409-13. doi: 10.1097/BSD.0b013e318201bf94. PMID 21150658
- [Result] Geck MJ, Eismont FJ. Surgical options for the treatment of cervical spondylotic myelopathy. Orthop Clin North Am. 2002 Apr;33(2):329-48. doi: 10.1016/s0030-5898(02)00002-0. PMID 12389279
- [Result] Komotar RJ, Mocco J, Kaiser MG. Surgical management of cervical myelopathy: indications and techniques for laminectomy and fusion. Spine J. 2006 Nov-Dec;6(6 Suppl):252S-267S. doi: 10.1016/j.spinee.2006.04.029. PMID 17097545
- [Result] Kadanka Z, Mares M, Bednanik J, Smrcka V, Krbec M, Stejskal L, Chaloupka R, Surelova D, Novotny O, Urbanek I, Dusek L. Approaches to spondylotic cervical myelopathy: conservative versus surgical results in a 3-year follow-up study. Spine (Phila Pa 1976). 2002 Oct 15;27(20):2205-10; discussion 2210-1. doi: 10.1097/01.BRS.0000029255.77224.BB. PMID 12394893
- [Result] Emery SE, Bohlman HH, Bolesta MJ, Jones PK. Anterior cervical decompression and arthrodesis for the treatment of cervical spondylotic myelopathy. Two to seventeen-year follow-up. J Bone Joint Surg Am. 1998 Jul;80(7):941-51. doi: 10.2106/00004623-199807000-00002. PMID 9697998
- [Result] Liu X, Min S, Zhang H, Zhou Z, Wang H, Jin A. Anterior corpectomy versus posterior laminoplasty for multilevel cervical myelopathy: a systematic review and meta-analysis. Eur Spine J. 2014 Feb;23(2):362-72. doi: 10.1007/s00586-013-3043-7. Epub 2013 Oct 5. PMID 24097230
- [Result] Rhee JM, Riew KD, Spivak JM, et al. Cervical spondylotic myelopathy: including ossification of the posterior longitudinal ligamented. Rosemont, IL, 2006.
- [Result] Malone A, Meldrum D, Bolger C. Gait impairment in cervical spondylotic myelopathy: comparison with age- and gender-matched healthy controls. Eur Spine J. 2012 Dec;21(12):2456-66. doi: 10.1007/s00586-012-2433-6. Epub 2012 Jul 24. PMID 22825630
- [Result] Kuhtz-Buschbeck JP, Johnk K, Mader S, Stolze H, Mehdorn M. Analysis of gait in cervical myelopathy. Gait Posture. 1999 Jul;9(3):184-9. doi: 10.1016/s0966-6362(99)00015-6. PMID 10575079
- [Result] Singh A, Choi D, Crockard A. Use of walking data in assessing operative results for cervical spondylotic myelopathy: long-term follow-up and comparison with controls. Spine (Phila Pa 1976). 2009 May 20;34(12):1296-300. doi: 10.1097/BRS.0b013e3181a09796. PMID 19412138
- [Result] Maezawa Y, Uchida K, Baba H. Gait analysis of spastic walking in patients with cervical compressive myelopathy. J Orthop Sci. 2001;6(5):378-84. doi: 10.1007/s007760170002. PMID 11845345
- [Result] Lee JH, Lee SH, Seo IS. The characteristics of gait disturbance and its relationship with posterior tibial somatosensory evoked potentials in patients with cervical myelopathy. Spine (Phila Pa 1976). 2011 Apr 15;36(8):E524-30. doi: 10.1097/BRS.0b013e3181f412d9. PMID 21224774
- [Result] Tetreault L, Goldstein CL, Arnold P, Harrop J, Hilibrand A, Nouri A, Fehlings MG. Degenerative Cervical Myelopathy: A Spectrum of Related Disorders Affecting the Aging Spine. Neurosurgery. 2015 Oct;77 Suppl 4:S51-67. doi: 10.1227/NEU.0000000000000951. PMID 26378358
- [Result] Creath R, Kiemel T, Horak F, Jeka JJ. The role of vestibular and somatosensory systems in intersegmental control of upright stance. J Vestib Res. 2008;18(1):39-49. PMID 18776597
- [Result] Wall PD, Noordenbos W. Sensory functions which remain in man after complete transection of dorsal columns. Brain. 1977 Dec;100(4):641-53. doi: 10.1093/brain/100.4.641. No abstract available. PMID 564735
- [Result] Ross RT. Dissociated loss of vibration, joint position and discriminatory tactile senses in disease of spinal cord and brain. Can J Neurol Sci. 1991 Aug;18(3):312-20. doi: 10.1017/s0317167100031875. PMID 1913366
- [Result] Takayama H, Muratsu H, Doita M, Harada T, Yoshiya S, Kurosaka M. Impaired joint proprioception in patients with cervical myelopathy. Spine (Phila Pa 1976). 2005 Jan 1;30(1):83-6. doi: 10.1097/00007632-200501010-00015. PMID 15626986
- [Result] Bohm PE, Fehlings MG, Kopjar B, Tetreault LA, Vaccaro AR, Anderson KK, Arnold PM. Psychometric properties of the 30-m walking test in patients with degenerative cervical myelopathy: results from two prospective multicenter cohort studies. Spine J. 2017 Feb;17(2):211-217. doi: 10.1016/j.spinee.2016.08.033. Epub 2016 Aug 31. PMID 27592193
- [Result] Tetreault L, Kopjar B, Cote P, Arnold P, Fehlings MG. A Clinical Prediction Rule for Functional Outcomes in Patients Undergoing Surgery for Degenerative Cervical Myelopathy: Analysis of an International Prospective Multicenter Data Set of 757 Subjects. J Bone Joint Surg Am. 2015 Dec 16;97(24):2038-46. doi: 10.2106/JBJS.O.00189. PMID 26677238
- [Result] Nouri A, Tetreault L, Singh A, Karadimas SK, Fehlings MG. Degenerative Cervical Myelopathy: Epidemiology, Genetics, and Pathogenesis. Spine (Phila Pa 1976). 2015 Jun 15;40(12):E675-93. doi: 10.1097/BRS.0000000000000913. PMID 25839387
- [Result] Dubousset J. Three-dimensional analysis of the scoliotic deformity. The pediatric spine: principles and practiceed. New York: Raven Press Ltd, 1994.
- [Result] Shumway-Cook A, Anson D, Haller S. Postural sway biofeedback: its effect on reestablishing stance stability in hemiplegic patients. Arch Phys Med Rehabil. 1988 Jun;69(6):395-400. PMID 3377664
- [Result] Haddas R, Lieberman IH. Correction to: A method to quantify the "cone of economy". Eur Spine J. 2018 May;27(5):1188. doi: 10.1007/s00586-018-5475-6. PMID 29396767
- [Result] Tanishima S, Nagashima H, Ishii H, Fukata S, Dokai T, Murakami T, Morio Y. Significance of Stabilometry for Assessing Postoperative Body Sway in Patients with Cervical Myelopathy. Asian Spine J. 2017 Oct;11(5):763-769. doi: 10.4184/asj.2017.11.5.763. Epub 2017 Oct 11. PMID 29093787
- [Result] Yoshikawa M, Doita M, Okamoto K, Manabe M, Sha N, Kurosaka M. Impaired postural stability in patients with cervical myelopathy: evaluation by computerized static stabilometry. Spine (Phila Pa 1976). 2008 Jun 15;33(14):E460-4. doi: 10.1097/BRS.0b013e318178e666. PMID 18552660
- [Result] Haddas R, Lieberman I, Arakal R, Boah A, Belanger T, Ju K. Effect of Cervical Decompression Surgery on Gait in Adult Cervical Spondylotic Myelopathy Patients. Clin Spine Surg. 2018 Dec;31(10):435-440. doi: 10.1097/BSD.0000000000000719. PMID 30222623
- [Result] Haddas R, Arakal R, Aghyarian S, et al. Gait Analysis on Adult Cervical Spondylotic Myelopathy Surgical Patients. 17th Annual Meeting of the International Society for the Advancement of Spine Surgery. Boca Raton, FL, USA, 2017.
- [Result] Haddas R, Arakal R, Aghyarian S, et al. Gait Analysis on Adult Cervical Spondylotic Myelopathy Surgical Patients. Orthopaedic Research Society 2017 annual meeting. San Diego, CA, 2017.
- [Result] Glantz SA. Primer of Biostatisticsed: McGraw-Hill Medical, 2011.